CLINICAL TRIAL: NCT03132727
Title: Interest of MRI in Preoperative Staging for the Laryngeal and Hypopharyngeal Cancer
Acronym: Larynx MRI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0632
Record Dates: First submitted 2017-03-29; First posted 2017-04-28 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Hypopharyngeal Carcinoma; Laryngeal Carcinoma
MeSH Terms: conditions — Hypopharyngeal Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pharyngo laryngeal MRI: Patient with a laryngeal or hypopharyngeal cancer at any stage, with a doubt about cartilage invasion and eligible for surgical treatment for which there is an indication for performing an MRI in addition to CT at the discretion of the investigator
  Interventions: Other: Pharyngo laryngeal MRI

INTERVENTIONS:
Other: Pharyngo laryngeal MRI — Patients will be outgoing a pharyngolaryngeal MRI, with injection of gadolinium, in addition to the CT imaging. They will have this MRI in case of doubt about cartilage invasion. It will be realised during the time between the CT imaging and the day of surgery.
  Device : gadolinium-based MRI contrast agent This will be realized according to the standard procedure.

SUMMARY:
To determine if MRI can detect preoperative invasion of cartilage by laryngeal and hypopharyngeal carcinoma, and to compare it to CT imaging and histopathology in excised larynges and/or hypopharynges.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old
* Patient with a laryngeal or hypopharyngeal cancer at any stage
* Patient eligible for a surgical treatment in multidisciplinary consultation
* Patient who did not oppose its participation to the study
* Indication for performing an MRI in addition to CT at the discretion of the investigator

Exclusion Criteria:

* Patient with an ASA ("American Society of Anesthesiologists", international anesthesia classification) score ≥ 3,
* Patient with a chirurgical contraindication
* Patient with a MRI contraindication
* Pregnant or nursing woman
* Adult requiring protection (guardianship, supervision)
* Patient participating in interventional research (Excluding physiological studies and interventional research involving only minimal risks and constraints that do not interfere with the analysis of the primary outcome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a laryngeal or hypopharyngeal cancer at any stage, with a doubt about cartilage invasion and eligible for surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Endoscopy | 1-4 weeks
  Tumor stage and cartilage invasion as determined by endoscopy : invaded/non invaded/undetermined
CT scan | 1-4 weeks
  Tumor stage and cartilage invasion as determined by CT scan : invaded/non invaded/undetermined
MRI | 1-4 weeks
  Tumor stage and cartilage invasion as determined by MRI : invaded/non invaded/undetermined
Anatomopathological analysis | 2-4 weeks
  Tumor stage and cartilage invasion as determined by histopathology in excised pieces : invaded/non invaded/undetermined

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CERUSE, Pr, Principal Investigator — Service ORL et chirurgie cervico-faciale, Hôpital de la Croix rousse
Locations (1):
- Service ORL et chirurgie cervico-faciale, Hôpital de la Croix rousse, Lyon, France